CLINICAL TRIAL: NCT01561963
Title: A Phase 1, Open-label, Three-period, Fixed-sequence Study to Evaluate the Effects of Rifampin on the Pharmacokinetics of Apremilast (CC-10004) in Healthy Subjects
Brief Title: A Drug-Drug Interaction Study to Evaluate the Effect of Rifampin on the Pharmacokinetics of Apremilast
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CC-10004-CP-025
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Results first posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Healthy Subjects
Keywords: Apremilast; drug interaction; pharmacokinetics
MeSH Terms: interventions — apremilast; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Apremilast and Rifampin (Experimental): Participants received the following 3 treatment regimens:
  * A single oral dose of 30 mg apremilast on Day 1 (Period 1);
  * A single oral dose of 30 mg apremilast followed 5 minutes later by a 30-minute intravenous infusion of 600 mg rifampin on Day 5 (Period 2);
  * Once daily oral doses of 600 mg rifampin for 15 days (from Day 7 to Day 21) with a single oral dose of 30 mg apremilast co-administered with the rifampin dose on Day 20 (Period 3).
  Interventions: Drug: Apremilast; Drug: Rifampin Oral Capsules; Drug: Rifampin IV Solution

INTERVENTIONS:
Drug: Apremilast — Tablets for oral administration
  Other Names: CC-10004; Otezla®
Drug: Rifampin Oral Capsules — Capsules for oral administration
  Other Names: RIFADIN™
Drug: Rifampin IV Solution — Intravenous (IV) solution
  Other Names: RIFADIN™

SUMMARY:
The purpose of this study is to evaluate how the pharmacokinetics of apremilast may be affected by a single intravenous dose of rifampin and multiple oral doses of rifampin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects of any ethnic origin between ages of 18 and 55 with a body mass index between 18 and 33

Exclusion Criteria:

* Recent history (i.e., within 3 years) of any clinically significant neurological, gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, endocrine, hematological, dermatological, psychological, allergic or other major disorders.
* Use of any prescribed or non-prescribed systemic or topical medication (including vitamins and herbal medicines, e.g. St. John's Wort) within 30 days of the first dose, unless an exception is granted by the sponsor.
* Presence of any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism, and excretion, or plans to have elective or medical procedures during the conduct of the trial.
* Exposure to an investigational drug (new chemical entity) within 30 days prior to the first dose administration

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2012-04-01 (Actual); Study Completion 2012-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Quintiles, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Liu Y, Zhou S, Wan Y, Wu A, Palmisano M. The impact of co-administration of ketoconazole and rifampicin on the pharmacokinetics of apremilast in healthy volunteers. Br J Clin Pharmacol. 2014 Nov;78(5):1050-7. doi: 10.1111/bcp.12448. PMID 24962564
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at one clinical site in Overland Park, Kansas, USA.
Groups:
- Apremilast and Rifampin: Participants received the following 3 treatment regimens:
  Period 1: A single oral dose of 30 mg apremilast on Day 1; Period 2: A single oral dose of 30 mg apremilast followed 5 minutes later by a 30-minute intravenous (IV) infusion of 600 mg rifampin on Day 5; Period 3: Once daily oral doses of 600 mg rifampin for 15 days (from Day 7 to Day 21) with a single oral dose of 30 mg apremilast co-administered with the rifampin dose on Day 20.
Period: Overall Study
Arm/Group | Apremilast and Rifampin
Started | 21
Received Period 1 Treatment | 21
Received Period 2 Treatment | 20
Received Period 3 Treatment | 20
Completed | 20
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Apremilast and Rifampin: Participants received the following 3 treatment regimens:
  Period 1: A single oral dose of 30 mg apremilast on Day 1; Period 2: A single oral dose of 30 mg apremilast followed 5 minutes later by a 30-minute intravenous infusion of 600 mg rifampin on Day 5; Period 3: Once daily oral doses of 600 mg rifampin for 15 days (from Day 7 to Day 21) with a single oral dose of 30 mg apremilast co-administered with the rifampin dose on Day 20.
Arm/Group | Apremilast and Rifampin
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12
  Black or African American | 9
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 29.14 (2.974)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUCt) of Apremilast
Description: Plasma concentrations of apremilast were determined by means of a validated, sensitive, and specific high performance liquid chromatography/tandem mass spectrometric (LC-MS/MS) assay.
Time Frame: Pre-dose and at 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36, and 48 hours following apremilast dosing on Days 1, 5, and 20
Population: The pharmacokinetic population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Apremilast Alone: Participants received a single oral dose of 30 mg apremilast on Day 1 (Period 1).
- Apremilast + IV Rifampin: Participants received a single oral dose of 30 mg apremilast followed 5 minutes later by a 30-minute intravenous infusion of 600 mg rifampin on Day 5 (Period 2).
- Apremilast + Multiple Dose Oral Rifampin: Participants received once daily oral doses of 600 mg rifampin for 15 days (from Day 7 to Day 21) with a single oral dose of 30 mg apremilast co-administered with the rifampin dose on Day 20 (Period 3).
Arm/Group | Apremilast Alone | Apremilast + IV Rifampin | Apremilast + Multiple Dose Oral Rifampin
Number analyzed (Participants) | 21 | 19 | 19
ng*h/mL | 3070 (31.3) | 2940 (31.3) | 850 (33.7)
Statistical Analysis 1: Comparison: Apremilast Alone vs Apremilast + IV Rifampin; The effect of rifampicin on the PK of apremilast was evaluated using a linear mixed effect analysis of variance on the log-transformed values of AUCt of apremilast, to estimate the mean ratio of apremilast administered with and without rifampicin treatment. The model included treatment as fixed effect, and subject as a random effect; Test type: Equivalence — No statistically significant interaction between apremilast and rifampicin was confirmed if both the upper and lower 90% confidence interval (CI) limits for the geometric least squares mean ratios of apremilast administered with rifampicin to apremilast alone fell within the no effect boundary of 80% to 125%; Ratio of Geometric Least Squares Means = 96.35, 90% CI 2-sided [88.56 to 104.82] — Apremilast + IV Rifampin / Apremilast Alone
Statistical Analysis 2: Comparison: Apremilast Alone vs Apremilast + Multiple Dose Oral Rifampin; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — No statistically significant interaction between apremilast and rifampicin was confirmed if both the upper and lower 90% CI limits for the geometric least squares mean ratios of apremilast administered with rifampicin to apremilast alone fell within the no effect boundary of 80% to 125%; Ratio of Geometric Least Squares Means = 27.88, 90% CI 2-sided [25.63 to 30.34] — Apremilast + Multiple Dose Oral Rifampin / Apremilast Alone

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC∞) of Apremilast
Description: as for outcome 1
Time Frame: Pre-dose and at 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36, and 48 hours following apremilast dosing on Days 1, 5, and 20
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Apremilast Alone | Apremilast + IV Rifampin | Apremilast + Multiple Dose Oral Rifampin
Number analyzed (Participants) | 21 | 19 | 19
ng*h/mL | 3120 (31.5) | 2980 (31.2) | 869 (32.9)
Statistical Analysis 1: Comparison: Apremilast Alone vs Apremilast + IV Rifampin; The effect of rifampicin on the PK of apremilast was evaluated using a linear mixed effect analysis of variance on the log-transformed values of AUC∞ of apremilast, to estimate the mean ratio of apremilast administered with and without rifampicin treatment. The model included treatment as fixed effect, and subject as a random effect; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Ratio of Geometric Least Squares Means = 95.71, 90% CI 2-sided [87.99 to 104.12] — Apremilast + IV Rifampin / Apremilast Alone
Statistical Analysis 2: Comparison: Apremilast Alone vs Apremilast + Multiple Dose Oral Rifampin; [analysis description as in outcome 2, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Ratio of Geometric Least Squares Means = 27.96, 90% CI 2-sided [25.70 to 30.41] — Apremilast + Multiple Dose Oral Rifampin / Apremilast Alone

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Apremilast
Description: as for outcome 1
Time Frame: Pre-dose and at 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36, and 48 hours following apremilast dosing on Days 1, 5, and 20
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Apremilast Alone | Apremilast + IV Rifampin | Apremilast + Multiple Dose Oral Rifampin
Number analyzed (Participants) | 21 | 19 | 19
ng/mL | 290 (24.5) | 331 (25.1) | 166 (23.2)
Statistical Analysis 1: Comparison: Apremilast Alone vs Apremilast + IV Rifampin; The effect of rifampicin on the PK of apremilast was evaluated using a linear mixed effect analysis of variance on the log-transformed values of Cmax of apremilast, to estimate the mean ratio of apremilast administered with and without rifampicin treatment. The model included treatment as fixed effect, and subject as a random effect; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Ratio of Geometric Least Squares Means = 113.07, 90% CI 2-sided [103.18 to 123.91] — Apremilast + IV Rifampin / Apremilast Alone
Statistical Analysis 2: Comparison: Apremilast Alone vs Apremilast + Multiple Dose Oral Rifampin; [analysis description as in outcome 3, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Ratio of Geometric Least Squares Means = 56.80, 90% CI 2-sided [51.84 to 62.25] — Apremilast + Multiple Dose Oral Rifampin / Apremilast Alone

4. Primary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of Apremilast
Description: as for outcome 1
Time Frame: Pre-dose and at 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36, and 48 hours following apremilast dosing on Days 1, 5, and 20
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Apremilast Alone | Apremilast + IV Rifampin | Apremilast + Multiple Dose Oral Rifampin
Number analyzed (Participants) | 21 | 19 | 19
hours | 2.00 [0.50 to 5.00] | 1.50 [0.50 to 5.00] | 1.00 [0.50 to 5.00]
Statistical Analysis 1: Comparison: Apremilast Alone vs Apremilast + IV Rifampin; Tmax was analyzed using nonparametric methods. The median difference and 90% CI of the median difference were calculated from the Hodges-Lehrmann estimate; Test type: Other; p = 0.2656, Wilcoxon signed rank test; Median Difference = -0.25, 90% CI 2-sided [-0.75 to 0.00] — Apremilast + IV Rifampin - Apremilast Alone
Statistical Analysis 2: Comparison: Apremilast Alone vs Apremilast + Multiple Dose Oral Rifampin; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.1141, Wilcoxon signed rank test; Median Difference = -0.50, 90% CI 2-sided [-1.00 to 0.00] — Apremilast + Multiple Dose Oral Rifampin - Apremilast Alone

5. Primary Outcome: Estimate of the Terminal Elimination Half-life (T1/2) of Apremilast in Plasma
Description: as for outcome 1
Time Frame: Pre-dose and at 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36, and 48 hours following apremilast dosing on Days 1, 5, and 20
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Apremilast Alone | Apremilast + IV Rifampin | Apremilast + Multiple Dose Oral Rifampin
Number analyzed (Participants) | 21 | 19 | 19
hours | 8.12 (14.1) | 7.35 (18.5) | 6.13 (24.8)

6. Primary Outcome: Apparent Total Plasma Clearance (CL/F) of Apremilast
Description: as for outcome 1
Time Frame: Pre-dose and at 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36, and 48 hours following apremilast dosing on Days 1, 5, and 20
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Apremilast Alone | Apremilast + IV Rifampin | Apremilast + Multiple Dose Oral Rifampin
Number analyzed (Participants) | 21 | 19 | 19
L/h | 9.60 (31.5) | 10.1 (31.2) | 34.5 (32.9)

7. Primary Outcome: Apparent Volume of Distribution (Vz/F) of Apremilast
Description: as for outcome 1
Time Frame: Pre-dose and at 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36, and 48 hours following apremilast dosing on Days 1, 5, and 20
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Apremilast Alone | Apremilast + IV Rifampin | Apremilast + Multiple Dose Oral Rifampin
Number analyzed (Participants) | 21 | 19 | 19
liters | 112 (35.8) | 107 (43.4) | 305 (51.6)

ADVERSE EVENTS:
Time Frame: Period 1 (Apremilast Alone): Day 1 to day 4; Period 2 (Apremilast + IV Rifampin): Day 5 to day 6; Period 3 (Apremilast + Multiple Dose Oral Rifampin): Day 7 up to day 32; Overall Study (All Treatment Regimens): Up to 32 days
Groups:
- Overall Study - All Treatment Regimens: Participants received the following 3 treatment regimens:
  Period 1: A single oral dose of 30 mg apremilast on Day 1; Period 2: A single oral dose of 30 mg apremilast followed 5 minutes later by a 30-minute intravenous infusion of 600 mg rifampin on Day 5; Period 3: Once daily oral doses of 600 mg rifampin for 15 days (from Day 7 to Day 21) with a single oral dose of 30 mg apremilast co-administered with the rifampin dose on Day 20.
Arm/Group | Apremilast Alone | Apremilast + IV Rifampin | Apremilast + Multiple Dose Oral Rifampin | Overall Study - All Treatment Regimens
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20 | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 2/21 | 4/20 | 9/20 | 12/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Apremilast Alone (N=21) | Apremilast + IV Rifampin (N=20) | Apremilast + Multiple Dose Oral Rifampin (N=20) | Overall Study - All Treatment Regimens (N=21)
CONJUNCTIVAL HYPERAEMIA (Eye disorders) | 0 | 1 | 0 | 1
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 | 0 | 1 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1 | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 1 | 1 | 1
DYSPHAGIA (Gastrointestinal disorders) | 0 | 0 | 1 | 1
ASTHENIA (General disorders) | 0 | 0 | 1 | 1
CHILLS (General disorders) | 0 | 0 | 1 | 1
FEELING HOT (General disorders) | 0 | 0 | 1 | 1
INFUSION SITE ERYTHEMA (General disorders) | 0 | 1 | 0 | 1
RHINITIS (Infections and infestations) | 0 | 0 | 2 | 2
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 | 0 | 1 | 1
HEPATIC ENZYME INCREASED (Investigations) | 0 | 0 | 1 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
MUSCLE TWITCHING (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
HEADACHE (Nervous system disorders) | 2 | 1 | 1 | 4
MUSCLE CONTRACTIONS INVOLUNTARY (Nervous system disorders) | 0 | 0 | 1 | 1
DYSURIA (Renal and urinary disorders) | 0 | 0 | 1 | 1
TESTICULAR PAIN (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.